CLINICAL TRIAL: NCT06520969
Title: Prevelance of Uterine Vein and Uterine Vein System Variations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Albayrak, MD, Gynecologic Oncology Fellow, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2248661
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Uterine Vein Injury Left; Uterine Vein Injury Right

STUDY DESIGN:
Intervention Model Description: Endometrium and cervical cancer patients that will be operated in Istanbul University School of Medicine, Dept. of Obstetrics and Gynecology, Division of Oncology will be included. Anatomic details such as the presence, number of superficial and deep uterine veins, calibers, anatomical relationships with hypogastric arteries and veins, ureters, vesicouterine ligaments will be described systematically and bilaterally for every consenting women after pelvic spaces are opened before pelvic lypmhadenectomy and hysterectomy. All regarding information will be photographed for every patient bilaterally and recorded on data sheet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prevalance and anatomical variations of superficial and deep veins (Other): Single arm anatomical study describing the prevalance and anatomical variations of superficial and deep veins in endometrial and cervical cancer patients
  Interventions: Other: Prevelance of Uterine Vein and Uterine Vein System Variations (anatomical study)

INTERVENTIONS:
Other: Prevelance of Uterine Vein and Uterine Vein System Variations (anatomical study) — Single arm anatomical study describing the prevalance and anatomical variations of superficial and deep veins in endometrial and cervical cancer patients
  Other Names: Single arm anatomical study describing the prevalance and anatomical variations of superficial and deep veins in endometrial and cervical cancer patients

SUMMARY:
Contrary to the uterine arterial system, our knowledge about superficial and deep uterine vein prevalence and anatomic variations are limited. The present study aims to deepen and clarify our knowledge on superficial and deep uterine vein anatomy, prevalence and relationship with other neighbouring structures which may be helpful in uterine transplantation and radical hysterectomy operations.

DETAILED DESCRIPTION:
Despite that two veins draining the uterus, superficial and deep, are described, their true anatomy, number, calibers, trajectories, relationships with sympathetic and parasympathetic nerves and internal iliac vasculature and ureters are quite limited. Additionally, variations of these vasculature are much less described. The aim of this study is to increase the our current knowledge about these anatomical information and also to calculate the prevalence of superficial and deep uterine veins which may potentially decrease the possible complications such as bleeding in uterine transplantation surgery and nerve sparing radical hysterectomy for cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

Endometrium and cervical cancer patients that will be operated -

Exclusion Criteria:

Any women in whom uterine vascular anatomy that might be changed for a specific disease such as myomas, uterine infections, etc.

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Endometrium and cervical cancer patients that will be operated
Enrollment: 100 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
To describe the prevalence of uterine vein and uterine vein system variations | 2 years
  To describe the prevalence of uterine vein and uterine vein system variations

CONTACTS AND LOCATIONS:
Overall Officials: Samet Topuz, MD, Study Director — Istanbul Univrsity
Locations (1):
- Istanbul University Medical Faculty Dept. of Obstet Gynecol, Division of Gynecologic Oncology, Istanbul, Istanbul / Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all information stated in this document is open to to third parties whitout any limitations
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: no time frame limit, all open for all times